CLINICAL TRIAL: NCT01249768
Title: Observational Study Assessing the Diagnostic Contribution of 3-Tesla MRI, CSF Analysis and a Second Opinion in a Specialized Movement Disorder Centre, in Differentiating Between Parkinson's Disease and Atypical Parkinsonism
Brief Title: Parkinson's Disease, Diagnostic Observations (PADDO)
Acronym: PADDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Marjolein Aerts, dr. M.B. Aerts, Radboud University Medical Center
Other Study IDs: PADDO
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson's Disease; Atypical Parkinsonism
Keywords: Prospective study; diagnostic accuracy; CSF; MRI
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, cerebrospinal fluids
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: The cohort will consist of 150 patients with a hypokinetic rigid syndrome and a disease duration of maximum 36 months

SUMMARY:
Background:

Parkinson's Disease and the Atypical Parkinsonian Disorder (like Multiple System Atrophy, Progressive Supranuclear Palsy, Corticobasal Degeneration, Lewy Body Dementia) are disease entities with partly common symptomatology. Especially very early in the course of disease, the differentiation between both disease entities can be challenging, even for specialists in the field of movement disorder. However, the establishment of a correct diagnosis is very important for adequate patientcounseling, treatment and the correct inclusion of patients in research trials. Ancillary diagnostic investigations are looked upon to aid in this diagnostic dilemma.

Objective:

To investigate the value of ancillary diagnostic investigations, more specific MRI, analysis of cerebrospinal fluids and a second opinion in a specialized movement disorder centre, to differentiate Parkinson's disease and the Atypical Parkisonisonian disorder.

ELIGIBILITY:
Inclusion Criteria:

* Hypokinetic rigid syndrome
* Disease duration of maximum 36 months

Exclusion Criteria:

* Probable diagnosis of PD without any red flags
* Probable diagnosis MSA
* Probable diagnosis PSP
* Diagnosis CBD
* Diagnosis DLB
* Probable diagnosis Vascular Parkinsonism
* Other neurodegenerative disease than parkinsonism
* A prior history of brain surgery
* Instable comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a hypokinetic-rigid syndrome with a disease duration of maximum 36 months and in whom a definitive diagnosis has not been established yet.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
percentage of correct diagnosis for each of the specified ancillary investigations | 36 months
  Percentage of correct diagnosis for each of the specified ancillary investigations to differentiate between either PD or atypical parkinsonism

SECONDARY OUTCOMES:
Percentage of correct diagnosis for each of the specified ancillary investigations | 36 months
  Percentage of correct diagnosis for each of the specified ancillary investigations(MRI, CSF analysis, and second opinion) to differentiate between the specific diagnosis (PD, MSA, PSP, CBD, LBD, VaP)

CONTACTS AND LOCATIONS:
Overall Officials: M Verbeek, PhD, MSc, Principal Investigator — Radboud University Medical Center; B Bloem, Prof, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] van Rumund A, Aerts MB, Esselink RAJ, Meijer FJA, Verbeek MM, Bloem BR. Parkinson's Disease Diagnostic Observations (PADDO): study rationale and design of a prospective cohort study for early differentiation of parkinsonism. BMC Neurol. 2018 May 16;18(1):69. doi: 10.1186/s12883-018-1072-x. PMID 29764386